CLINICAL TRIAL: NCT00809393
Title: Comparison of Two Tranexamic Acid Dose Regimens on Transfusion Needs During Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Dose-ranging Study of Two Doses of Tranexamic Acid During Cardiac Surgery
Acronym: Exacylcardio
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008/27
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Cardiopulmonary Bypass; Hemorrhage
Keywords: Antifibrinolytic; Tranexamic acid; Cardiopulmonary bypass; Transfusion; Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low dose (Active Comparator): low dose tranexamic acid
  Interventions: Drug: tranexamic acid
- high dose (Experimental)
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — 10 mg/kg
  Arms: low dose
Drug: tranexamic acid — 30 mg/kg
  Arms: high dose

SUMMARY:
Cardiac surgery with CardioPulmonary Bypass (CPB) exposes to per and postoperative bleeding, and may lead to allogenic blood transfusion re-intervention and many adverse outcomes. Prophylactic use of tranexamic Acid (TA) has been shown to decrease blood loss and blood transfusion during cardiac surgery.There currently are multiple dosing regimens for TA for cardiac surgery.Preliminary dose-response study has shown that low prophylactic dose of TA would be as accurate for haemostatic efficacy as higher dose.

The primary objective of this tri-center, prospective, double-blinded, randomised trial is to compare two administrations and dosing regimens of TA during cardiac surgery with CPB on the perioperative blood loss.

In addition to the clinical study, a pharmacokinétic/pharmacodynamic study will be conducted.

Patients are divided in two groups: low and high risk surgery. Methods: After written informed consent, patients are randomly assigned to one of the two treatment groups. The low dose TA group is: 10 mg/kg TA given over 15 min, followed by an infusion of 1 mg/kg/h throughout the operation, and 1 mg/kg into the CPB prime volume. The high dose group is :30 mg/kg TA given over 15 min, followed by an infusion of 16 mg/kg/h throughout the operation, and 2 mg/kg into the CPB prime volume. Hemodynamic and anaesthesia care will be as usual. A blood salvage device will be systematically used. The triggers for transfusion will be: red blood cells: haemoglobin less than 8 g/dl or 6 g/dl during CBP; Plasma: PT less than 50% or INR more than 1.5; platelets: platelets count less than 50/70 G/mm3; fibrinogen: fibrinogen less than 1g/l . All patients will receive standard anaesthesia and perioperative care.

In 60 consecutive patients in the principal investigator center, 5 blood samples will allow to assess the plasmatic concentration of tranexamic acid at different time of the surgery procedure:

1. Baseline
2. 5 min after the loading dose
3. 10 min after the beginning of bypass
4. at the discontinuation of the infusion
5. 1 hour after the discontinuation Plasmatic dosage will be assessed using a high performance liquid chromatography technique.

Patients will be stratified in two groups for the statistical analysis; low and high risk surgery. Analysis will be in intention to treat. 300 patients should be recruited in each group to detect an absolute difference of respectively 10% (low risk cardiac surgery) and 20% (high risk cardiac surgery) in the number of patients exposed to allogenic blood transfusion between patients receiving high dose TA regimen and those receiving low dose TA regimen, assuming a power of 80% and a two-tailed value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Any type of cardiac surgical procedure requiring CPB (including coronary artery bypass grafting, valve repair or replacement, aortic surgery, endocarditis).

Exclusion Criteria:

* Emergency surgery, age < 18 years old, pregnancy, history of allergy to TA, history of seizure or thromboembolism event, history of previous antifibrinolytic or thrombolytic therapy within 5 days of surgery, coagulation disorder, liver disease, renal failure (clearance < 30 ml/min), Jehovah witness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary study outcome is the number of patients in each group exposed to allogenic blood transfusion during the first 7 days after surgery. | 7th day

SECONDARY OUTCOMES:
Number of fresh plasma frozen units, platelets units needed for the 7 days , post operative blood loss in the 24 hours, needed or repeat surgery due to haemorrhage for the 24 hours following surgery, in-hospital death at 7 and 28 days. | 28th day
Relationship between blood loss during the first 24 hours following the surgery and plasmatic concentration of acid tranexamic | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - department of anaesthesiology, CHU Jean Minjoz, Besançon
  - department of anesthesiology, Haut Leveque Hospital, Bordeaux
  - department of anesthesiology, Bichat Hospital, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Grassin-Delyle S, Tremey B, Abe E, Fischler M, Alvarez JC, Devillier P, Urien S. Population pharmacokinetics of tranexamic acid in adults undergoing cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2013 Dec;111(6):916-24. doi: 10.1093/bja/aet255. Epub 2013 Jul 23. PMID 23880099